CLINICAL TRIAL: NCT03683368
Title: Extended Wear of a Steel and a Teflon Insulin Infusion Set
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mylife Diabetes Care AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YPU105
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft cannula first (Experimental): Subjects will be randomized (50%) to the soft cannula infusion set for two weeks and then will be switched to the steel needle infusion set for two additional weeks. Participants will aim for 7 day use of each infusion set type twice, starting with the soft cannula infusion set.
  Interventions: Device: YpsoPump Orbit soft; Device: YpsoPump Orbit micro
- Steel cannula first (Experimental): Subjects will be randomized (50%) to the steel cannula infusion set for two weeks and then will be switched to the soft cannula infusion set for two additional weeks. Participants will aim for 7 day use of each infusion set type twice, starting with the steel cannula infusion set.
  Interventions: Device: YpsoPump Orbit soft; Device: YpsoPump Orbit micro

INTERVENTIONS:
Device: YpsoPump Orbit soft — Insulin infusion sets will be used for up to 7 days or until failure
Device: YpsoPump Orbit micro — Insulin infusion sets will be used for up to 7 days or until failure

SUMMARY:
This is a cross-over study to evaluate if insulin infusion sets can be used up to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least 12 months
* Using an insulin pump for at least 12 months
* Age ≥18 years
* Hemoglobin A1c level less than or equal to 8.5%
* Willing to use mylife™ YpsoPump® system while they are participating in the study
* Willing to use NovoRapid® insulin while they are participating in the study
* An understanding of and willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

* Diabetic ketoacidosis in the past 3 months prior to enrollment
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 3 months prior to enrollment
* Urea, Creatinine, ALT more than three times the upper limit of normal, or thrombocytopenia (<150 G/l)
* Female subjects: pregnancy, lactation period, lack of a negative pregnancy test (except in case of menopause, sterilization or hysterectomy), or unwilling to use an acceptable form of contraception during the study (for sexually active subjects of childbearing potential)
* Known severe tape reactions or allergies
* Known severe nickel allergies
* History of frequent catheter abscesses associated with pump therapy
* Serious acute or chronic disease besides diabetes mellitus or an anamnesis which might, in the opinion of the investigator, pose a risk to the subject, e.g. seizure disorder, adrenal disorder, dialysis for renal failure, cystic fibrosis, active infection
* Any incapacity or general condition that, in the opinion of the investigator, prevents adequate compliance with the study procedures, e.g. mental or visual incapacity, language barriers, alcohol or drug misuse
* Dependency from the sponsor or the clinical investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Time to infusion set failure due to an occlusion | up to 7 days
  an occlusion is defined by blood ketone concentration is > or = 0.6 mmol/l with blood glucose (BG) concentration >250 mg/dl, or BG concentration is >250 mg/dl for more than 2 h and a subsequent correction bolus failed, or pump occlusion alarm that cannot be fixed.

SECONDARY OUTCOMES:
Frequency of early infusion set changes | up to 7 days
Time to early infusion set changes | up to 7 days
Frequency of early infusion set changes due to infusion site infection | up to 7 days
Median infusion set wearing time | up to 7 days
Daily mean glucose | day 1, 2, 3, 4, 5, 6, 7
  Based on Continuous Glucose Monitoring
Daily mean glucose | day 1, 2, 3, 4, 5, 6, 7
  Based on self measured blood glucose
Total daily insulin dose | day 1, 2, 3, 4, 5, 6, 7
Glucose variability | day 1, 2, 3, 4, 5, 6, 7
  Coefficient of variation

CONTACTS AND LOCATIONS:
Overall Officials: Guido Freckmann, MD, Principal Investigator — Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm; Andreas Buhr, Dr., Study Director — Ypsomed AG, Burgdorf, Switzerland
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No